CLINICAL TRIAL: NCT04878562
Title: Improving Chicago Older Adult Opioid and Pain Management Through Patient-Centered Clinical Decision Support and Project ECHO
Brief Title: I-COPE Study: Opioid Use and Pain Management in Older Adults
Acronym: I-COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); ACCESS Community Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB20-1580
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain; Opioids; Opioid-use Disorder
Keywords: older adults; electronic health record; chronic pain; opioid use disorder
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: We will conduct a nonhybrid pragmatic implementation-effectiveness stepped wedge cluster-randomized study in which clinics will be the randomized clusters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-COPE Intervention (Experimental): 5 out of the 25 participating primary care sites are randomly assigned to any of the 5 steps. The ICOPE intervention is implemented after a pre interventional period of 3-15 months. The intervention is implemented during 8 weeks. The length of the post interventional period is 11-23 months.
  Interventions: Behavioral: I-COPE
- No intervention (No Intervention): Standard of care offered to all patients.

INTERVENTIONS:
Behavioral: I-COPE — The patient survey will be sent out via MyChart 3 days before the visit. It asks about current pain, goals, treatment history, treatment preferences, and health status. Alternatively, patients will be asked to compete a survey in clinic on paper or a tablet. The surveys will be identical, except screening for screening for depression and opioid use will depend on the availability of previous scores. Survey and the EHR will help auto-generate best practice advisories (BPAs) and a tailored smart set. The smartset is based on AGS and CDC guidelines for chronic pain and opioids. It shows which treatment options are not recommended based on the patient's history, comorbidities, and preferences. The smartset also includes links to decision aid and patient education tools. Personalized action plan will be created with pain rating and goal, treatment plan, and relevant tips and educational materials. Action plan will be clearly laid out using max 6 grade reading level, and simple graphics.
  Arms: I-COPE Intervention

SUMMARY:
Adults over 65 years of age are at higher risk of experiencing chronic pain and adverse events from opioids and opioid use disorder (OUD). Older adults are more likely to inadequately report their pain due to age-related health, which may lead to undertreatment of pain. In the last two decades, opioid prescriptions to treat chronic pain among older adults increased at a rate of nine times what it was previously. This surge is accompanied with a drastic increase of older adults visiting emergency departments due to opioid abuse, misuse, overdose, and addictions to heroin and cocaine. In consequence, chronic pain, opioids, and OUD have become a major crisis in the United States among older adults. The I-COPE program is an intervention that offers providers a set of smart tools for a more effective and efficient geriatric pain, opioid, and OUD management. The aim of the I-COPE program is to evaluate integration of shared decision-making, patient-centered clinical decision support tools, and Project ECHO® to address the critical need to integrate effective treatment for older adults with chronic pain, opioid use, and OUD. Patient-centered clinical decision support (PCCDS) tools provide clinicians with information presented at the right time and tailored to the individual patient, improving communications, care, and patient-provider satisfaction. Shared decision making (SDM) is a highly effective collaborative framework when there are many choices and there is uncertainty about the optimal treatment choice. Project ECHO® is a tested model for delivery of subspecialized medical knowledge to community clinicians. The research into these strategies is supported by the Agency for Healthcare Research and Quality (AHRQ) through the opioid action plan (OAP) initiative. Based on the survey responses the PCCDS will develop a list of pain treatments that are preferable for older adults to use, based on their individual histories. From the PCCDS, an individualized patient action plan will be generated. The action plan will be clearly laid out, use patient-centered language at an ≤ 6th grade level, and simple graphics. It will feature the patient-reported overall goal, current pain rating and pain goal, as well as provide information on changes made to the chronic pain treatment plan. Information about signs of opioid side effects, misuse and opioid overdoses will be included for patients who are taking opioids, as well as instructions for naloxone administration.

DETAILED DESCRIPTION:
I-COPE program intervention includes four components: patient survey, geriatric PCCDS tool, patient action plan, and provider education.

Patient survey. Three days before each of their scheduled PCP visits, patients will be asked to complete a survey during electronic check-in. If patients have not completed the questionnaire when they arrive on the day of their appointment, they will be asked by the patient services representatives to complete it in the waiting area on paper or using a tablet, or by the medical assistant to complete it during patient triage. In addition to the I-COPE survey patients will be screened for depression and drug abuse. Medical assistants will be trained to enter their responses into the EHR. A caregiver may help the patient complete the questionnaire. Responses will be saved in the patient's medical record and accessible to their care team.

Geriatric PCCDS tool. Information from the patient questionnaire and the EHR will be used to automatically generate a passive alert (best practice advisory) and a tailored smart set which PCPs can open during the visit. The alert will be triggered if a patient responds that they want to discuss pain at their visit or if they screen positive for a possible substance use disorder. The PCCDS was designed with a set of decision rules based on AGS and CDC guidelines for chronic pain and opioids. The PCCDS tool features five sections: All patients (self-management strategies), Oral non-opioid medications, Acute-on-chronic pain only, Opioid medications, and OUD treatment. The PCCDS shows which treatment options are recommended, not recommended, or contraindicated based on the patient's history, comorbidities, and preferences. For instance, if a patient screens positive for depression the Antidepressants smartgroup within the Oral non-opioid medications section will be open and labelled as recommended. Alternative versions of other smartgroups exist for patients with chronic kidney disease of various stages, presence of certain medication, and results of the drug abuse screening. The PCCDS tool also includes links to a conversation tool and patient self-management education tools. The PCCDS tool may be accessed by a provider in cases where patient did not complete the survey.

Patient action plan. At the end of the visit, a personalized action plan will be generated for patients featuring their pain rating and goal, the treatment plan they agreed upon with their PCP, and relevant educational materials. The action plan will be clearly laid out using patient-centered language, maximum 6th grade reading level, and simple graphics. It will be printed out as a part of the after-visit summary.

Provider education. PCPs may opt into an intensive Project ECHO course that offers more geriatric clinical content and EHR updates with real-word cases. Project ECHO (Extension for Community Health Outcomes) is an innovative workforce development model for expanding primary care capacity in underserved communities. It uses videoconferencing technology to "telementor" community-based clinicians via didactic education, group problem solving with actual cases brought by clinicians, and expert advice on implementing best practices. Project ECHO® is possibly a cost-effective strategy for improving clinician competence and behaviors, while likely improving patient outcomes. The curriculum will be delivered in 8-weekly hour-long sessions. Each session will include didactic topics delivered by an interdisciplinary team of content experts, and two 15-minute problem-solving exercises using real-world cases brought by participating PCPs. PCPs will review how they can use the I-COPE Program toolkit with each case. Didactic content will include a walkthrough of the PCCDS and education on the demographics of pain and OUD, special considerations for pain management (e.g., cognitive impairment, functional impairment, social determinants, and caregivers), principles of SDM and assessing patient preferences, pharmacology and pain medications, non-pharmacologic pain management options, and recognition and management of OUD. The abridged version of the ECHO training will be made available online for PCPs to access on their own time if needed.

ELIGIBILITY:
Inclusion Criteria:

* age over 65 years AND
* receives care at a participating clinical site AND
* history of chronic pain AND/OR
* opioid prescription in the last 28 days AND/OR
* history of opioid use disorder AND/OR

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with high initial pain scores (≥6) who experience a 30% reduction in scores | 6 months
  Percentage of patients with high initial pain scores (≥6) who experience a 30% reduction in scores
Increase diversity of recommended pain treatments | 6 months
  More types of treatment are represented in patient's treatment plan. In I-COPE smartset pain treatments are grouped into 4 types: self-management, referrals to specialists, non-opioid medications, and opioid medications.
Decrease higher-risk pain treatments | 6 months
  Discontinuation of opioid/Beer's Criteria medications or decrease in daily milligram equivalents of opioid/Beer's Criteria medications.

SECONDARY OUTCOMES:
Change in pain scores among older adults with and without chronic pain diagnoses and high initial pain scores | 6 months
  Change in pain scores among older adults with and without chronic pain diagnoses and high initial pain scores
Increase in guideline concordant opioid prescriptions | 6 months
  Increase in naloxone prescribing in patients with >50mg equivalents of opioids or OUD; Increase in the number of annual drug screens in patient with chronic opioid use; Decrease in co-prescribing of opioids and benzodiazepines
Decrease in percentage of patients prescribed each high-risk treatments | 6 months
  High-risk treatments are defined as opioids and Beer's criteria medications
Increase in percentage of patients prescribed each low-risk treatments | 6 months
  Low-risk treatments include all pain treatments except opioids and Beer's criteria medications.
Percentage of eligible patients who receive an I-COPE action plan | 6 months
  Percentage of eligible patients who receive an I-COPE action plan
Percentage of physicians who use the I-COPE program | 6 months
  Percentage of physicians in study sites who use the I-COPE program
Percentage of clinics who use the I-COPE program | 6 months
  Percentage of clinics who successfully implement the I-COPE program

CONTACTS AND LOCATIONS:
Overall Officials: Mim Ari, MD, Principal Investigator — University of Chicago; Neda Laiteerapong, MD, Principal Investigator — University of Chicago; Katherine Thompson, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago Medicine, Chicago, Illinois
  - Access Community Health Network, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
This is a clinic-level intervention study. Research team will only receive a limited data set with no individual participant data.

REFERENCES:
- [Background] Gianni W, Ceci M, Bustacchini S, Corsonello A, Abbatecola AM, Brancati AM, Assisi A, Scuteri A, Cipriani L, Lattanzio F. Opioids for the treatment of chronic non-cancer pain in older people. Drugs Aging. 2009 Dec;26 Suppl 1:63-73. doi: 10.2165/11534670-000000000-00000. PMID 20136170
- [Background] American Geriatrics Society Panel on Pharmacological Management of Persistent Pain in Older Persons. Pharmacological management of persistent pain in older persons. J Am Geriatr Soc. 2009 Aug;57(8):1331-46. doi: 10.1111/j.1532-5415.2009.02376.x. Epub 2009 Jul 2. No abstract available. PMID 19573219
- [Background] Abdulla A, Adams N, Bone M, Elliott AM, Gaffin J, Jones D, Knaggs R, Martin D, Sampson L, Schofield P; British Geriatric Society. Guidance on the management of pain in older people. Age Ageing. 2013 Mar;42 Suppl 1:i1-57. doi: 10.1093/ageing/afs200. PMID 23420266
- [Background] Guerriero F. Guidance on opioids prescribing for the management of persistent non-cancer pain in older adults. World J Clin Cases. 2017 Mar 16;5(3):73-81. doi: 10.12998/wjcc.v5.i3.73. PMID 28352631
- [Background] West NA, Severtson SG, Green JL, Dart RC. Trends in abuse and misuse of prescription opioids among older adults. Drug Alcohol Depend. 2015 Apr 1;149:117-21. doi: 10.1016/j.drugalcdep.2015.01.027. Epub 2015 Jan 31. PMID 25678441
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Lewis ET, Cucciare MA, Trafton JA. What do patients do with unused opioid medications? Clin J Pain. 2014 Aug;30(8):654-62. doi: 10.1097/01.ajp.0000435447.96642.f4. PMID 24281287
- [Background] Wu LT, Blazer DG. Illicit and nonmedical drug use among older adults: a review. J Aging Health. 2011 Apr;23(3):481-504. doi: 10.1177/0898264310386224. Epub 2010 Nov 17. PMID 21084724
- [Background] Huhn AS, Strain EC, Tompkins DA, Dunn KE. A hidden aspect of the U.S. opioid crisis: Rise in first-time treatment admissions for older adults with opioid use disorder. Drug Alcohol Depend. 2018 Dec 1;193:142-147. doi: 10.1016/j.drugalcdep.2018.10.002. Epub 2018 Oct 18. PMID 30384321
- [Background] Carter MW, Yang BK, Davenport M, Kabel A. Increasing Rates of Opioid Misuse Among Older Adults Visiting Emergency Departments. Innov Aging. 2019 Mar 7;3(1):igz002. doi: 10.1093/geroni/igz002. eCollection 2019 Jan. PMID 30863796
- [Background] Kuerbis A, Sacco P, Blazer DG, Moore AA. Substance abuse among older adults. Clin Geriatr Med. 2014 Aug;30(3):629-54. doi: 10.1016/j.cger.2014.04.008. Epub 2014 Jun 12. PMID 25037298
- [Background] Schultz SK, Arndt S, Liesveld J. Locations of facilities with special programs for older substance abuse clients in the US. Int J Geriatr Psychiatry. 2003 Sep;18(9):839-43. doi: 10.1002/gps.994. PMID 12949852
- [Derived] Kagarmanova A, Sparkman H, Laiteerapong N, Thompson K, Rosul L, Lazar D, Staab E, Wan W, Kass A, Ari M. Improving the management of chronic pain, opioid use, and opioid use disorder in older adults: study protocol for I-COPE study. Trials. 2022 Jul 27;23(1):602. doi: 10.1186/s13063-022-06537-w. PMID 35897111